CLINICAL TRIAL: NCT03935841
Title: Metabolic Differences of an Oral and Intravenous Dose of 3-hydroxybutyrate (3-OHB).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Nikolaj Fibiger Rittig, Principal investigator, MD, PhD, and clinical researcher, University of Aarhus
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1-10-72-56-19
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Healthy; Incretin Effect; Ketosis
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-OHB orally (Experimental): 36 gram 3-OHB salt consumed orally
  Interventions: Dietary Supplement: 3-OHB salt (NaCl)
- 3-OHB intravenously (Active Comparator): Variable amounts of 3-OHB salt given i order to replicate the same individual plasma concentrations measured during the experimental arm.
  Interventions: Dietary Supplement: 3-OHB salt (NaCl)

INTERVENTIONS:
Dietary Supplement: 3-OHB salt (NaCl) — 36 gram 3-OHB salt diluted in 500 ml sterile water

SUMMARY:
An open-labeled intervention study testing healthy, lean, and male volunteers on two separate occasions:

1. blood sampling after consuming 36 gram 3-Hydroxybutyrate (3-OHB) salt.
2. blood sampling while given a variable rate of 3-OHB salt intravenously to replicate the concentrations seen during oral consumption.

The primary outcome is differences in insulin concentrations (incremental AUC) 180 minutes after 3-OHB consumed orally vs. intravenously.

Secondary outcomes includes iAUC for other gastrointestinal hormones and substrates (Glucagon, GLP-1, GIP, glucose, and 3-OHB) Gastric emptying will be evaluated using 1500 mg Paracetamol consumption before each intervention day. Urine will be analyzed for ketone concentrations/excretion rates.

DETAILED DESCRIPTION:
An open-labeled intervention study testing healthy, lean, and male volunteers on two separate occasions with at least 48 hours apart.

1. blood sampling after consuming 36 gram 3-Hydroxybutyrate (3-OHB) salt.
2. blood sampling while given a variable rate of 3-OHB salt intravenously to replicate the concentrations seen during oral consumption.

The primary outcome is differences in insulin concentrations (incremental AUC) 180 minutes after 3-OHB consumed orally vs. intravenously.

Secondary outcomes includes iAUC for other gastrointestinal hormones and substrates (Glucagon, GLP-1, GIP, glucose, and 3-OHB) Gastric emptying will be evaluated using 1500 mg Paracetamol consumption before each intervention day. Urine will be analyzed for ketone concentrations/excretion rates.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* 19<BMI<30
* written og oral consent
* No allergies to paracetamol

Exclusion Criteria:

* Chronic disease or daily medical treatment
* Daily intake of ketones or ketogenic diets
* Speaks and understands Danish
* Screening blood sample abnormalities

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
plasma insulin | 180 minutes
  incremental area under the curve (iAUC) for plasma insulin concentrations {pmol/l}

SECONDARY OUTCOMES:
Plasma Glucagon | 180 minutes
  iAUC and concentrations of (Glucagon {pg/ml}
Gastric emptying | 180 minutes
  Paracetamol test, 1500 mg following interventions and measuring plasma paracetamol {micromol/l}
Urine 3-OHB | 180 minutes
  Excretion rates {gram/hour} will be estimated as = urine output {L} x urine 3-OHB concentration {mmol/l} x 0.1041 {g/mmol}/180 minutes
Plasma GLP1 | 180 minutes
  iAUC and concentrations of GLP-1 {pmol/l},
Plasma GIP | 180 minutes
  iAUC and concentrations of GIP {pmol/l},
Plasma glucose | 180 minutes
  iAUC and concentrations of glucose {mmol/l},
Plasma free fatty acids | 180 minutes
  iAUC and concentrations of free fatty acids {mmol/l},
Plasma 3-OHB | 180 minutes
  iAUC and concentrations of 3-OHB {mmol/l})
Plasma Ghrelin | 180 minutes
  iAUC and concentrations of Ghrelin {ng/l})
Plasma PYY | 180 minutes
  iAUC and concentrations of PYY {pg/ml})
height | at time 0 minutes
  height {meters}
weight | at time 0 minutes
  weight {kg}
BMI | time 0 minutes
  Body mass index = weight/height^2
Blood pressure | time 0 minutes and 180 minutes
  Arm blood pressure
Satiety questionnaire (Blundell et al. 2010) | At 0, 60, 120, and 180 minutes
  VAS/NRS-score of hunger, fullness, satiety, desire, and prospective consumption
Ad libitum food intake | at time = 180 minutes
  gram (and kcal) intake of an ad libitum meal (sandwich)

CONTACTS AND LOCATIONS:
Overall Officials: Niels Jessen, Professor, Study Director — Aarhus University Hospital
Locations (1):
- Department of Diabetes and Hormone Diseases (DoH), Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersen MGB, Lauritzen ES, Svart MV, Stoy J, Sondergaard E, Thomsen HH, Kampmann U, Bjerre M, Jessen N, Moller N, Rittig N. Nutrient sensing: LEAP2 concentration in response to fasting, glucose, lactate, and beta-hydroxybutyrate in healthy young males. Am J Clin Nutr. 2023 Dec;118(6):1091-1098. doi: 10.1016/j.ajcnut.2023.10.007. Epub 2023 Oct 14. PMID 37844838
- [Derived] Rittig N, Svart M, Thomsen HH, Vestergaard ET, Rehfeld JF, Hartmann B, Holst JJ, Johannsen M, Moller N, Jessen N. Oral D/L-3-Hydroxybutyrate Stimulates Cholecystokinin and Insulin Secretion and Slows Gastric Emptying in Healthy Males. J Clin Endocrinol Metab. 2020 Oct 1;105(10):dgaa483. doi: 10.1210/clinem/dgaa483. PMID 32717058